CLINICAL TRIAL: NCT04254315
Title: OPTIMA: Psychological Distress and the Effect of Intensive Group Based Cognitive Therapy in Patients With Newly Diagnosed Ischemic Heart Disease: A Randomised Controlled Trial Protocol
Brief Title: OPTIMA: Psychological Distress and the Effect of Intensive Group Based Cognitive Therapy in Patients With Newly Diagnosed Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Hanne Kruuse Rasmusen, Associate Professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-16042832
Record Dates: First submitted 2020-01-18; First posted 2020-02-05 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Heart Disease; Heart Valve Diseases; Psychological Distress
Keywords: Group based cognitive therapy; Ischemic Heart Disease; Heart Valve Diseases; Psychological Distress
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: A randomized study with
  * Intervention group
  * Control group with psychological distress
  * Control group without psychological distress (not part of randomization)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cardiac rehabilitation+cognitive therapy (Experimental): The intervention group receives usual cardiac rehabilitation, which consists of 8-wk supervised outpatient exercise with 2 weekly sessions of 1,5 hr with high-intensity interval and resistance training. The program was complemented with a weekly session of group-based patient education for 1,5 hr on heart disease, psychological issues and diet counseling. In addition, patients had one or more individual sessions with a cardiologist and a nurse respectively.
  In addition, the intervention group follows a standardized group based cognitive therapy program with participation of maximum four patients, consisting of 5 sessions (each 2 hours) performed by a trained cardiac rehabilitation nurse.
  Interventions: Behavioral: Group based cognitive therapy
- Cardiac rehabilitation (No Intervention): The control group receives usual cardiac rehabilitation, which consists of 8-wk supervised outpatient exercise with 2 weekly sessions of 1,5 hr with high-intensity interval and resistance training. The program was complemented with a weekly session of group-based patient education for 1,5 hr on heart disease, psychological issues and diet counseling. In addition, patients had one or more individual sessions with a cardiologist and a nurse respectively. .
- Control group without psychological distress (No Intervention): The control group receives usual cardiac rehabilitation, which consists of 8-wk supervised outpatient exercise with 2 weekly sessions of 1,5 hr with high-intensity interval and resistance training. The program was complemented with a weekly session of group-based patient education for 1,5 hr on heart disease, psychological issues and diet counseling. In addition, patients had one or more individual sessions with a cardiologist and a nurse respectively. .

INTERVENTIONS:
Behavioral: Group based cognitive therapy — Patients are informed about the Optima program in the inclusion interview, and patients are participating in groups of maximum 4 persons. Each of the 5 session has a duration of 1,5 - 2 hours.
  The psychologist have developed the content of each session, with attention to thoughts and feelings regarding the current situation after a heart-condition, and the effects on life conditions. Patients get the tools to overcoming the difficulties, they experience, f.x. anxiety and stress.
  When other hospitals are joining the Optima project, the project nurse and psychologist are training the hospital staff as well as supervising.
  Arms: Cardiac rehabilitation+cognitive therapy

SUMMARY:
The overall objectives of the Optima project is to: (1) Compare the effect of standardized group based cognitive therapy and cardiac rehabilitation versus usual cardiac rehabilitation in patients with sign of psychological distress measured by a questionnaire (HADS score), (2) To investigate spontaneous variation in psychological distress with HADS over time in order to optimize time of measuring HADS. (3) To investigate if the intervention can be implemented to other cardiac rehabilitation sites with the same effect as on BFH (that it is not person dependent).

DETAILED DESCRIPTION:
HYPOTHESIS: There will be a significant difference in anxiety and depression score between intervention and usual care groups after intervention, in favor of the intervention group.

METHODS: Optima is a multi-center, prospective, randomized clinical trial in patients with newly diagnosed ischemic heart disease (IHD) or heart valve replacement, and concomitant significant score of psychological distress using the Hospital Anxiety and Depression Score (HADS) (HADS A(Anxiety) /D(Depression) ≥8 or HADS>15), age <65 years. Patients with HADS D≥11 and Beck Depression Inventory (BDI)>17 are evaluated by psychiatrists to offer the best treatment. 148 patients will be randomized to either intervention or control group. All patients are offered usual cardiac rehabilitation, and in addition, the intervention group is offered standardized group based cognitive therapy with the participation of maximum four patients, consisting of 5 sessions (each 2 hours) performed by a trained cardiac rehabilitation nurse. The intervention was developed on experiences from a Liaison nurse, who offered up to five individual consultations to patients with psychological distress. Together with a psychologist specialized in cognitive therapy the investigators developed a program based on cognitive behavioral methods from cognitive therapy as well as Acceptance and commitment therapy (ACT). Each session consists of specific cognitive models, which the patient can use in everyday life.

INTERVENTION: Patients are informed about the Optima program in the inclusion interview, and patients are participating in groups of maximum 4 persons. Each of the 5 session has a duration of 1,5 - 2 hours.

The psychologist have developed the content of each session, with attention to thoughts and feelings regarding the current situation after a heart-condition, and the effects on life conditions. Patients get the tools to overcoming the difficulties, they experience, f.x. anxiety and stress.

When other hospitals are joining the Optima project, the project nurse and psychologist are training the hospital staff as well as supervising.

The session are planned as follows Session 1: Identifying your values

* What is important in my life?
* How has my heart-condition effected my life?
* Where do I want to be in my life? And what challenges it? Session 2: Anxiety and techniques to reduce anxiety
* What is anxiety?
* Anxiety and heart symptoms
* Circle of anxiety
* Techniques to reduce anxiety, relaxation and breathing Session 3: Consequences of own behavior and behavioral analysis
* Behavior that reduces self-expression
* Heart disease and behavior
* Consequences of own behavior Session 4: Concerns and strategies for dealing with them
* What are concerns?
* The Worry Tree and how to use it.
* Strategies for handling concerns. Session 5: The balance between demands and capacity
* Thoughts about the future
* Working life, relations and family

Sessions are followed up with two interviews after 3 and 6 months, where the following are assessed:

* The Hospital Anxiety and Depression Scale (HADS) score
* Heart-related Quality of Life (HeartQoL)
* Blood samples
* Clinical assessment: Functional Classification of Angina (CCS), New York Heart Association (NYHA) score, Blood pressure, medical status, smoking/nonsmoking, weight, physical activity (self-assessment) cardiovascular readmissions
* Employment status
* return to work
* present psychosocial status

QUESTIONNAIRES: Questionnaires include validated assessment tools:

HADS: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire that assesses anxiety and depression level in medically ill persons who are not admitted in psychiatric wards. The scale range is from 0 to 42, the lesser the score, the lesser signs of psychological distress. The scale offers two scores, HADS-A and HADS-D, and consists of seven questions to assess anxiety and seven questions to assess depression.

HeartQol: Heart-related Quality of Life is a disease-specific questionnaire that measures health-related quality of life in patients with heart disease. The questionnaire consists of 14 items and provides two subscales: a 10-item physical subscale and a 4-item emotional subscale, which are scored from 0 to 3. Higher scores indicating better HRQL.

Also, a questionnaire that measures present psychosocial status/situation is used. The questionnaire is based on clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* HADS score > 8 for HADS-A or HADS-D
* Age < 65 years
* Able to speak and understand Danish

Exclusion Criteria:

* Participation in rehabilitation program within the last 2 years
* Ejection Fraction (EF) < 35%
* Other serious comorbidity that are expected to have a serious impact on life expectancy
* Known abuse of alcohol or euphoric drugs. Known more serious psychopathology such as schizophrenia, bipolar disorder, severe personality disorder, and treatment with psychoactive drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the RCT is anxiety and depression measured by HADS | 3 months follow-up
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire that assesses anxiety and depression level in medically ill persons who are not admitted in psychiatric wards. The scale range is from 0 to 42, the lesser the score, the lesser signs of psychological distress.The scale offers two scores, HADS-A and HADS-D, and consists of seven questions to assess anxiety and seven questions to assess depression.
The primary outcome of the RCT is anxiety and depression measured by HADS | 6 months follow-up
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire that assesses anxiety and depression level in medically ill persons who are not admitted in psychiatric wards. The scale range is from 0 to 42, the lesser the score, the lesser signs of psychological distress.The scale offers two scores, HADS-A and HADS-D, and consists of seven questions to assess anxiety and seven questions to assess depression.

SECONDARY OUTCOMES:
Adherence to cardiac rehabilitation, health-related quality of life measured by HeartQoL | 3 months follow-up
  Heart-related Quality of Life (HeartQoL) is a disease-specific questionnaire that measures health-related quality of life in patients with heart disease. The questionnaire consists of 14 items and provides two subscales: a 10-item physical subscale and a 4-item emotional subscale, which are scored from 0 to 3. Higher scores indicating better HRQL.Return to work, adherence to life style interventions, and cardiovascular readmissions. A questionnaire that measures present psychosocial status/situation. The questionnaire is based on clinical experience.
Adherence to cardiac rehabilitation, health-related quality of life measured by HeartQoL | 6 months follow-up
  Heart-related Quality of Life (HeartQoL) is a disease-specific questionnaire that measures health-related quality of life in patients with heart disease. The questionnaire consists of 14 items and provides two subscales: a 10-item physical subscale and a 4-item emotional subscale, which are scored from 0 to 3. Higher scores indicating better HRQL.Return to work, adherence to life style interventions, and cardiovascular readmissions. A questionnaire that measures present psychosocial status/situation. The questionnaire is based on clinical experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology department, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Background] Damen NL, Versteeg H, Boersma E, Serruys PW, van Geuns RJ, Denollet J, van Domburg RT, Pedersen SS. Depression is independently associated with 7-year mortality in patients treated with percutaneous coronary intervention: results from the RESEARCH registry. Int J Cardiol. 2013 Sep 10;167(6):2496-501. doi: 10.1016/j.ijcard.2012.04.028. Epub 2012 May 3. PMID 22560933
- [Background] van Dijk MR, Utens EM, Dulfer K, Al-Qezweny MN, van Geuns RJ, Daemen J, van Domburg RT. Depression and anxiety symptoms as predictors of mortality in PCI patients at 10 years of follow-up. Eur J Prev Cardiol. 2016 Mar;23(5):552-8. doi: 10.1177/2047487315571889. Epub 2015 Feb 9. PMID 25665581
- [Background] Gulliksson M, Burell G, Vessby B, Lundin L, Toss H, Svardsudd K. Randomized controlled trial of cognitive behavioral therapy vs standard treatment to prevent recurrent cardiovascular events in patients with coronary heart disease: Secondary Prevention in Uppsala Primary Health Care project (SUPRIM). Arch Intern Med. 2011 Jan 24;171(2):134-40. doi: 10.1001/archinternmed.2010.510. PMID 21263103
- [Background] Blumenthal JA, Sherwood A, Smith PJ, Watkins L, Mabe S, Kraus WE, Ingle K, Miller P, Hinderliter A. Enhancing Cardiac Rehabilitation With Stress Management Training: A Randomized, Clinical Efficacy Trial. Circulation. 2016 Apr 5;133(14):1341-50. doi: 10.1161/CIRCULATIONAHA.115.018926. Epub 2016 Mar 21. PMID 27045127
- [Background] Zheng X, Zheng Y, Ma J, Zhang M, Zhang Y, Liu X, Chen L, Yang Q, Sun Y, Wu J, Yu B. Effect of exercise-based cardiac rehabilitation on anxiety and depression in patients with myocardial infarction: A systematic review and meta-analysis. Heart Lung. 2019 Jan;48(1):1-7. doi: 10.1016/j.hrtlng.2018.09.011. Epub 2018 Oct 23. PMID 30366575
- [Derived] Holdgaard A, Eckhardt-Hansen C, Lund T, Lassen CF, Sibiliz KL, Hofsten DE, Prescott E, Rasmusen HK. Intensive group-based cognitive therapy in patients with cardiac disease and psychological distress-a randomized controlled trial protocol. Trials. 2021 Jul 16;22(1):455. doi: 10.1186/s13063-021-05405-3. PMID 34271952